CLINICAL TRIAL: NCT04455568
Title: Establish a Telecare Model of Acute Coronary Syndrome Patient With Heart Stent Implantation by a Non-invasive Wearable Device and Artificial Intelligence Cloud System to Heart Failure Monitoring and Reducing Medical Adverse Events.
Brief Title: Establish a Telecare Model of Acute Coronary Syndrome Patient With Heart Stent Implantation by a Non-invasive Wearable Device and Artificial Intelligence Cloud to Reducing Medical Adverse Events.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Taipei Medical University WanFang Hospital (Other); Taipei Medical University Hospital (Other); Taipei Medical University (Other); Lotung Poh-Ai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: N202004123
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-06

CONDITIONS: Acute Coronary Syndrome; Percutaneous Transluminal Coronary Angioplasty
Keywords: Artificial Intelligence; Non-invasive Wearable Device; Telecare Model of Patient,; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Control Groups

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: Non-invasive Wearable Device, use ECG Wisdom bracelet
  Interventions: Device: use EKG Wisdom bracelet

INTERVENTIONS:
Device: use EKG Wisdom bracelet — Non-invasive Wearable Device (use EKG Wisdom bracelet)
  Other Names: control group (routine medical)

SUMMARY:
Heart disease is still one of the world's most important health problems, and it ranks second among the top ten causes of death among Taiwan. The main cause of death is acute coronary syndrome, and vascular stent placement is the main treatment method for acute coronary syndrome. The probability of restenosis in patients within half a year after a general stent is as high as 25% to 40%. Re-hospitalization and surgery is a big burden on patients and the country's medical costs. However, a set of convenient and accurate clinical tools to determine the prognosis of patients has not yet been developed. Miniaturized wearable devices have been the mainstream trend in medical development in recent years. ECG and heart sound analysis technology are an easy to used medical device for automatically calculating the parameters including EMAT (electromechanical activation time), S4, S4, SDI (Systolic dyssynchrony index). ECG and heart sound could evaluate the heart function, and has the potential to be an effective tools for prognosis and treatment guidelines. Heart rate variability (HRV) and Accelerationplethysmogram (APG) is also proved the predictive effect the outcome of patients.

This study is start on June 1 2020. We will enroll 400 patients who diagnosis of acute coronary syndrome and have been a heart stent surgery, and registry there medical history,routine examination and medication, ECG and heart, HRV and APG record at admission, pre-discharge and every routine return visit within I year after discharge.Patients will also wear ECG and PPG (Photoplethysmography) band ever day after discharge, and collected the longitutinal data .All subjects will be tracked the medical adverse events in 1 years after discharge, and compare the characteristic and prognosis value of between patients with and without events. Therefore, our purpose of this study is to drive an effective outcome prediction model by non-invasive device, and establish a telecare model of patient with heart stent implantation to reducing medical adverse events.

DETAILED DESCRIPTION:
This study is open, prospective study, multi-center, randomized controlled trial, unobtrusive research. This study is start on June 1 2020. We will enroll 400 patients who diagnosis of acute coronary syndrome and have been a heart stent surgery. And random allocation 200 experimental group (Non-invasive Wearable Device) and 200 control group (routine medical).

Ask whether the patients who meet the exclusion criteria are willing to participate in the screening (Screening), if they are willing to join and sign the consent of the subject, and after the patient's condition is stable, conduct an electrocardiogram (V0) before discharge from the hospital. On day 7 (±2 weeks), day 84 (±4 weeks), 168 days (±4 weeks), 252 days (±4 weeks), 336 days (±8 weeks) during routine clinical referral (V1-V5) Both are done once. The results of these two tests and other basic information of the patient, including Demography, Vital Signs, High, Weight, Medication, and European and Taiwan Cardiology Association recommended routine test results of high-risk patients, including Blood Chemistry Panel, NT-proBNP, Echocardiography, Myocardial Perfusion Scan, etc., will record the information of the logged-in subjects on the paper case report form. The CRF (case report form) only displays the study number, and no subject is available. In addition to the examination of each return visit, the subjects also took the ECG bracelet home at the time of discharge (V0) and wore it every day. After the discharge, the ECG was measured every morning and evening, and their personal activity and sleep were collected. Relevant information. After the subject was discharged from the hospital, the subject tracked the date of all adverse events due to cardiovascular disease within one year, including: heart failure, restenosis due to blood vessel, and non-fatal myocardial infarction , To do blood vessel-related surgery again, and data on the occurrence of death.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20-year-old
2. Patients performing general metal stent surgery
3. Diagnosis of Acute Coronary Syndrome
4. Willing to sign the consent form of the subject and cooperate with the return visit
5. Those who are admitted to the hospital and enter the general ward can receive the first ECG heart sound examination

Exclusion Criteria:

1. <20-year-old
2. Before the stent was installed, the same blood vessel had been used in patients with PCI (percutaneous coronary intervention) and CABG (Coronary artery bypass graft).
3. Those who cannot perform the first examination after being admitted to the hospital and entering the general ward
4. It is impossible to measure the group of ECG and heart sounds. For example, when using Pacemaker, the ECG showed ventricular tachycardia (VT) and Dextrocardia on admission.
5. Patients who are bedridden and have difficulty in cooperating with return visits
6. Any subject that the physician believes is at high risk for future uncooperative tracking
7. Direct participants in this program

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll 400 patients who diagnosis of acute coronary syndrome and have been a heart stent surgery. And random allocation 200 experimental group (Non-invasive Wearable Device) and 200 control group (routine medical).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
death | Within a year
  death
Restenosis | Within a year
  Restenosis
heart failure | Within a year
  heart failure

SECONDARY OUTCOMES:
heart disease re-hospitalization | Within a year
  heart disease re-hospitalization
Stroke re-hospitalization | Within a year
  Stroke re-hospitalization
Arrhythmia re-hospitalization | Within a year
  Arrhythmia re-hospitalization
Physician adjusts medicine | Within a year
  Physician adjusts medicine
Physician arranges examination early | Within a year
  Physician arranges examination early
Medical Compliance | Within a year
  Judged by the physician, when the patient returns to the consultation, the patient is asked about the compliance with the drug in the past, divided into presence and absence
Medical Costs | Within a year
  The sum of all medical and health insurance expenses of the patient in the past year

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Chi Liu, MD, Principal Investigator — Chief, Internal of Medicine

IPD SHARING:
Plan to Share IPD: Undecided